CLINICAL TRIAL: NCT01246700
Title: Sensory Attention Focused Exercise in Parkinson's Disease: A Randomized Double-Crossover Trial.
Brief Title: Sensory Attention Focused Exercise in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Life Financial Movement Disorders Research and Rehabilitation Centre (Other)
Collaborators: Canada, Young Men's Christian Association (YMCA) (Unknown); Parkinson Society Canada (Other); Canada, Sun Life Financial (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Quincy Almeida; Director of Sun Life Financial Movement Disorders Research and Rehabilitation Centre, Sun Life Financial Movement Disorders Research and Rehabilitation Centre; Wilfrid Laurier University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 225510
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Randomized single-blind crossover trial; Sensory Attention Focused Exercise
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Participants received 12 weeks of Sensory Attention Focused Exercise, then received 12 weeks of no exercise.
  Interventions: Other: Sensory Attention Focused Exercise (SAFEx)
- Group B (Experimental): Participants received no treatment for 12 weeks, then received Sensory Attention Focused Exercise for 12 weeks.
  Interventions: Other: Sensory Attention Focused Exercise (SAFEx)

INTERVENTIONS:
Other: Sensory Attention Focused Exercise (SAFEx) — Consisted of 12 weeks for SAFEx intervention, 3 times a week for an hour each session. Participants complete dynamic balance activities and a variety of seated stretches and range of motion activities. Participants are cued to focus on sensation and proprioception of limbs.
  Group A received SAFEx for 12 weeks then received no treatment for 12 weeks.
  Arms: Group A
Other: Sensory Attention Focused Exercise (SAFEx) — Consisted of 12 weeks for SAFEx intervention, 3 times a week for an hour each session. Participants complete dynamic balance activities and a variety of seated stretches and range of motion activities. Participants are cued to focus on sensation and proprioception of limbs.
  Group B received no treatment for 12 weeks, then received SAFEx for 12 weeks.
  Arms: Group B

SUMMARY:
The purpose of this study is 1.) to determine if sensory attention focused exercise is an effective management strategy for Parkinson's disease, and 2.) to identify if the benefits are a result of strength gains.

DETAILED DESCRIPTION:
Currently, there is no cure for Parkinson's disease (PD) and although medication offers symptom reduction, there are many negative side effects associated with medication use. Thus, there has been an increased emphasis on exercise interventions for symptom reduction. Recent research has shown that both sensory attention focused exercise (SAFEx) and strength training interventions improved disease severity more so than other exercise interventions (such as aerobic, aquatic and no exercise). Upon closer examination, SAFEx showed further symptom improvements than the strength training program. Thus exists the need to further examine SAFEx using a standardized protocol - a single-blind randomized double-crossover trial - that has been used sparingly in exercise interventions. In addition, the 30-second chair stand has been implemented into the testing protocol, as it has been shown to be a reliable measurement of functional strength for older adults. This test was implemented in order to identify the functional strength gains, if any, that are associated with SAFEx. It is hypothesized that the SAFEx intervention will improve disease symptoms in PD, and that the results will not be due to strength gains.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PD by a clinician/neurologist
* absence of mentation
* established medication schedule and dosage

Exclusion Criteria:

* mentation
* change in medication during period of study
* change in exercise level during period of study
* inability to complete the exercise program
* absence of 5 or more classes, or absence of 3 or more classes in sequence

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) III (motor score) | Baseline, 12 weeks and 24 weeks
  Assessment of patient's disease severity, completed by a blinded certified clinician.

SECONDARY OUTCOMES:
Timed up and go | Baseline, 12 weeks and 24 weeks
  Participants stand out of a chair, walk 3 meters, turn around and sit back down. This task is timed.
30 second chair stand | Baseline, 12 weeks and 24 weeks
  Participants instructed to stand from a seated position as many times as possible in 30 seconds. Number of completed stands is recorded.
Unified Parkinson's Disease Rating Scale (UPDRS) - I and II (self report of mentation, depression, and activities of daily living). | Baseline, 12 weeks and 24 weeks
  Participants complete a self-report questionnaire, and rank how they are feeling.
Grooved Pegboard | Baseline, 12 weeks and 24 weeks
  Participants must place and remove 25 pegs as fast as possible using a standard Grooved Pegboard. Participants are timed.
Step Length | Baseline, 12 weeks and 24 weeks
  Measured using GAITRite software.
Velocity | Baseline, 12 weeks and 24 weeks
  Assessed using GAITRite software.
Step to Step Length Variability | Baseline, 12 weeks and 24 weeks
  Assessed using GAITRite software.

CONTACTS AND LOCATIONS:
Overall Officials: Quincy J Almeida, Ph.D, Study Director — Sun Life Financial Movement Disorders Research and Rehabilitation Centre
Locations (1):
- Sun Life Financial Movement Disorders Research and Rehabilitation Centre, Waterloo, Ontario, Canada

REFERENCES:
- [Background] Sage MD, Almeida QJ. Symptom and gait changes after sensory attention focused exercise vs aerobic training in Parkinson's disease. Mov Disord. 2009 Jun 15;24(8):1132-8. doi: 10.1002/mds.22469. PMID 19373930
- [Background] Sage MD, Almeida QJ. A positive influence of vision on motor symptoms during sensory attention focused exercise for Parkinson's disease. Mov Disord. 2010 Jan 15;25(1):64-9. doi: 10.1002/mds.22886. PMID 19938164
- [Background] Nieuwboer A, Kwakkel G, Rochester L, Jones D, van Wegen E, Willems AM, Chavret F, Hetherington V, Baker K, Lim I. Cueing training in the home improves gait-related mobility in Parkinson's disease: the RESCUE trial. J Neurol Neurosurg Psychiatry. 2007 Feb;78(2):134-40. doi: 10.1136/jnnp.200X.097923. PMID 17229744
- [Background] Comella CL, Stebbins GT, Brown-Toms N, Goetz CG. Physical therapy and Parkinson's disease: a controlled clinical trial. Neurology. 1994 Mar;44(3 Pt 1):376-8. doi: 10.1212/wnl.44.3_part_1.376. PMID 8145901
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- See also: The Sun Life Movement Disorders Research and Rehabilitation Centre, based out of Wilfrid Laurier University, facilitates relevant research on Parkinson's disease. — http://www.wlu.ca/homepage.php?grp_id=2234